CLINICAL TRIAL: NCT07135492
Title: Intraoperative Continuous Noninvasive Hemoglobin Monitoring in Patients Undergoing Thoracic Surgery
Acronym: noninvasive Hb
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mona Mohamed Mogahed, Associate professor of Anesthesia, Tanta University
Other Study IDs: A01890
Record Dates: First submitted 2025-07-04; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Thoracic Anesthesia
Keywords: Thoracic; surgery; hemoglobin; transcutaneous oximetry.

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: continuous noninvasive hemoglobin monitoring — noninvasive hemoglobin monitoring, Rainbow® Adult ReSposable™ sensors (Rev E) were placed on either the ring or middle fingertip of each participant and connected to a Radical-7 Pulse CO-Oximeter (SET version 7601; Masimo Corp., Irvine, CA).

SUMMARY:
This study investigates the correlation between noninvasive hemoglobin monitoring (SpHb) and invasive hemoglobin measurement (InvHb) in guiding blood transfusions during thoracic surgeries.

Methods: A non-interventional design was used to evaluate the relationship between SpHb and InvHb readings in the context of transfusion decisions. Data were obtained from 80 patients aged 18 years or older undergoing thoracic procedures. Continuous SpHb monitoring was performed, and concurrent InvHb samples were collected for comparison. The primary endpoint was the degree of correlation between SpHb and InvHb values.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years and older who were subjected to open thoracic surgery
* the length of surgery was ≥ 4 hours

Exclusion Criteria:

* dysrhythmia
* coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients were monitored using ASA standard monitors, along with invasive arterial and/or central venous monitoring as part of their standard care.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2024-07-03 (Actual); Primary Completion 2025-07-03 (Actual); Study Completion 2025-07-04 (Actual)

PRIMARY OUTCOMES:
the correlation between continuous hemoglobin and inasive hemoglubin at the preoperative period | 6 Hours
  continuous hemoglobin % monitoring, Rainbow adult ReSposable™ sensors (rev E) were attached to the ring or middle fingertip of each subject and connected to a Radical-7 Pulse CO-Oximeter (SET version 7601; Masimo Corporation, Irvine, CA).
  invasive hemoglubin % monitoring, Blood samples were collected and analyzed using a satellite blood analyzer (Gem Premier 4000)
the correlation between continuous hemoglobin and inasive hemoglubin 1 hour after start of surgery | 6 Hours
  continuous hemoglobin % monitoring, Rainbow adult ReSposable™ sensors (rev E) were attached to the ring or middle fingertip of each subject and connected to a Radical-7 Pulse CO-Oximeter (SET version 7601; Masimo Corporation, Irvine, CA).
  invasive hemoglubin % monitoring, Blood samples were collected and analyzed using a satellite blood analyzer (Gem Premier 4000)
the correlation between continuous hemoglobin and inasive hemoglubin 2 hours after start of surgery | 6 Hours
  continuous hemoglobin % monitoring, Rainbow adult ReSposable™ sensors (rev E) were attached to the ring or middle fingertip of each subject and connected to a Radical-7 Pulse CO-Oximeter (SET version 7601; Masimo Corporation, Irvine, CA).
  invasive hemoglubin % monitoring, Blood samples were collected and analyzed using a satellite blood analyzer (Gem Premier 4000)
the correlation between continuous hemoglobin and inasive hemoglubin 3 hours after start of surgery | 6 Hours
  continuous hemoglobin % monitoring, Rainbow adult ReSposable™ sensors (rev E) were attached to the ring or middle fingertip of each subject and connected to a Radical-7 Pulse CO-Oximeter (SET version 7601; Masimo Corporation, Irvine, CA).
  invasive hemoglubin % monitoring, Blood samples were collected and analyzed using a satellite blood analyzer (Gem Premier 4000)
the correlation between continuous hemoglobin and inasive hemoglubin 4 hours after start of surgery | 6 Hours
  continuous hemoglobin % monitoring, Rainbow adult ReSposable™ sensors (rev E) were attached to the ring or middle fingertip of each subject and connected to a Radical-7 Pulse CO-Oximeter (SET version 7601; Masimo Corporation, Irvine, CA).
  invasive hemoglubin % monitoring, Blood samples were collected and analyzed using a satellite blood analyzer (Gem Premier 4000)
the correlation between continuous hemoglobin and inasive hemoglubin at the end of surgery | 6 Hours
  continuous hemoglobin % monitoring, Rainbow adult ReSposable™ sensors (rev E) were attached to the ring or middle fingertip of each subject and connected to a Radical-7 Pulse CO-Oximeter (SET version 7601; Masimo Corporation, Irvine, CA).
  invasive hemoglubin % monitoring, Blood samples were collected and analyzed using a satellite blood analyzer (Gem Premier 4000)
the correlation between continuous hemoglobin and inasive hemoglubin after recovery of the patient | 6 Hours
  continuous hemoglobin % monitoring, Rainbow adult ReSposable™ sensors (rev E) were attached to the ring or middle fingertip of each subject and connected to a Radical-7 Pulse CO-Oximeter (SET version 7601; Masimo Corporation, Irvine, CA).
  invasive hemoglubin % monitoring, Blood samples were collected and analyzed using a satellite blood analyzer (Gem Premier 4000)

CONTACTS AND LOCATIONS:
Locations (1):
- Ministry of health, Jeddah, Mekkah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Joseph B, Haider A, Rhee P. Non-invasive hemoglobin monitoring. Int J Surg. 2016 Sep;33(Pt B):254-257. doi: 10.1016/j.ijsu.2015.11.048. Epub 2015 Nov 30. PMID 26654895

DOCUMENTS (1):
  • Study Protocol (2024-07-13): https://cdn.clinicaltrials.gov/large-docs/92/NCT07135492/Prot_000.pdf